CLINICAL TRIAL: NCT01048710
Title: Treatment of Medial Compartmental Osteoarthritis Grade 1-4 (Kellgren-Lawrence) or Osteonecrosis With TomoFix™ Small or Conservatively
Brief Title: Treatment of Medial Compartmental Osteoarthritis Grade 1-4 With TomoFix™ Small or Conservatively
Status: Completed | Type: Observational
Sponsor: Synthes GmbH (Industry)
Collaborators: Johnson & Johnson K.K. Medical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: Tomofix_small
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis, Knee; Osteonecrosis
Keywords: Knee osteoarthritis; knee osteonecrosis; osteotomy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tomofix_small: Surgical treatment using TomoFix TM Small
  Interventions: Other: No intervention
- Conservative treatment: In the control group, patients who refused to have surgery will be allowed to be treated using different options of conservative treatment. The frequency of applications depends on the hospital and will therefore be documented in the study. An arthroscopy is not obligatory under this treatment group, but is permitted.
  The following conservative treatment methods are allowed:
  1. Physical therapy
  2. Specific exercises for the muscles
  3. Injections into the knee joint
  4. Brace
  5. Medication
  6. No therapy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The primary objective of this prospective multicenter study is to assess whether the functional outcome measured with the Knee Injury and Osteoarthritis Outcome Score (KOOS) for patients with medial unicompartmental osteoarthritis and osteonecrosis of the knee treated with open wedge high tibial osteotomy (HTO) using the TomoFix™ Small is better than the functional outcome after conservative treatment.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee (gonarthrosis) is a common medical condition and causes pain and disability. By 65 years of age, the majority of the US population has radiographic evidence of OA and 11% have symptomatic OA of the knee. In Japan, OA of the knee is more common due to the common sitting style with maximally flexed knees and parallel position of both legs.

High Tibial Osteotomy (HTO) for knee OA is a standard procedure in orthopedic surgery. Six years ago, HTO using TomoFix™ was introduced. Because Asian people have different geometric dimensions of the tibiae, an adaptation of size and shape was necessary, and the new TomoFix™ Small was developed. Although there is widespread literature concerning osteotomy for treating knee OA, literature assessing patient outcome after open wedge HTO using TomoFix™ is rare and for TomoFix™ Small, this data is still nonexistent. Therefore, the primary aim of the present multicenter study is to evaluate patient functional outcome using the KOOS. Since a proportion of patients with the indication for HTO refuse surgery and opt to receive conservative treatment, the functional results of patients treated with HTO using TomoFix™ Small will be compared with these patients.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age and older
* Patients with OA Grade 1-4 (Kellgren-Lawrence) or osteonecrosis (ON) Stage 2-4 (according to the Koshino classification)
* Indication for open wedge HTO with the TomoFix™ Small
* No ligamental laxity
* Signed written informed consent (by the subjects or legal guardian) and agreement to attend all planned follow-ups
* Willing and able to comply with the postoperative management program
* Able to understand and read country national language at an elementary level

Exclusion Criteria:

* Femoro-tibial angle (FTA) > 185o (standing view x-ray)
* Flexion contracture > 15o
* Total knee replacement or unicompartmental knee on the contralateral side
* Infections located between the middle of the femur and the ankle
* Systemic bacterial infections
* Severe osteoarthritis or surgery of the hip joint
* Smoking of more than 20 cigarettes per day
* Immunodeficiency or compromised host
* Patients who have participated in any other device or drug related clinical trial within the previous month
* ACL/PCL reconstruction of the same knee
* Severe osteoarthritis of the ipsilateral ankle joint

For conservative group only:

* HTO on the contralateral side
* Major surgery on both knees (minor surgery as arthroscopic meniscectomy and synovectomy is allowed)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Indication for open wedge HTO with the TomoFix™ Small presenting in the orthopaedic department of the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1 month, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, and 5 years

SECONDARY OUTCOMES:
Patient-evaluated function of the knee and quality of life, a. assessed with the Oxford-12-item knee score b. assessed with the WOMAC (as calculated from the KOOS) | 1 month, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, and 5 years
Clinician-evaluated function of the knee, assessed with the Japanese Orthopaedic Association (JOA) score | 1 month, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, and 5 years
Health-related quality of life assessed by the generic Short Form-36 (SF-36) instrument | 1 month, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, and 5 years
Range of motion (ROM) | 1 month, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, and 5 years
Local and general pain, assessed with the Visual Analogue Scale (VAS) | 1 month, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, and 5 years
Possibility and duration of the Japanese sitting style | 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, and 5 years
Surgery details, Postoperative treatment, Postoperative rehabilitation, Utilization | postoperative period
Evaluation of degenerated and regenerated cartilage (arthroscopic findings assessed according to ICRS and Outerbridge / Koshino) | intraoperative and after 2 years
Radiological parameters (e.g. union, delayed union, Kellgren-Lawrence classification, joint space narrowing, tibial slope, tibia vara, patella height according to Blackburne-Peel, modified Insall-Salvati ratio, subluxation of patella) | 1 month, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, and 5 years
Complications and mortality | 1 month, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Sawaguchi, MD, Principal Investigator — Toyama Municipal Hospital
Locations (1):
- Toyama Municipal Hospital, Toyama, Japan

REFERENCES:
- [Background] Takeuchi R, Aratake M, Bito H, Saito I, Kumagai K, Hayashi R, Sasaki Y, Akamatsu Y, Ishikawa H, Amakado E, Aota Y, Saito T. Clinical results and radiographical evaluation of opening wedge high tibial osteotomy for spontaneous osteonecrosis of the knee. Knee Surg Sports Traumatol Arthrosc. 2009 Apr;17(4):361-8. doi: 10.1007/s00167-008-0698-4. Epub 2009 Jan 23. PMID 19165468
- [Background] Takeuchi R, Ishikawa H, Aratake M, Bito H, Saito I, Kumagai K, Akamatsu Y, Saito T. Medial opening wedge high tibial osteotomy with early full weight bearing. Arthroscopy. 2009 Jan;25(1):46-53. doi: 10.1016/j.arthro.2008.08.015. Epub 2008 Oct 10. PMID 19111218
- [Background] Takeuchi R, Saito T, Koshino T. Clinical results of a valgus high tibial osteotomy for the treatment of osteoarthritis of the knee and the ipsilateral ankle. Knee. 2008 Jun;15(3):196-200. doi: 10.1016/j.knee.2008.02.002. Epub 2008 Mar 25. PMID 18367399